CLINICAL TRIAL: NCT01106547
Title: The Effect of a Preoperative Single-dose Methylprednisolone on the Postoperative Rehabilitation After Abdominal Hysterectomy: A Prospective, Double Blinded, Placebo Controlled Study
Brief Title: The Effect of a Preoperative Single-dose Methylprednisolone on the Postoperative Rehabilitation After Abdominal Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Anna Aabakke, Anna Aabakke, M.D., Holbaek Sygehus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Hysterektomistudiet; SJ-127 (Other: The Danish National Committee on Biomedical Research Ethics); 2010-018448-15 (EudraCT Number)
Record Dates: First submitted 2010-04-14; First posted 2010-04-20 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Hysterectomy; Methylprednisolone; Postoperative Pain
Keywords: abdominal hysterectomy; glucocorticoids; rehabilitation; postoperative pain; analgetics
MeSH Terms: conditions — Pain, Postoperative | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methylprednisolone (Experimental)
  Interventions: Drug: Methylprednisolone 125mg
- placebo/sodium chloride (Placebo Comparator)
  Interventions: Drug: Sodium Chloride 2 ml

INTERVENTIONS:
Drug: Methylprednisolone 125mg — Single dose 60-90 minutes preoperatively
  Other Names: Solu-medrol
  Arms: Methylprednisolone
Drug: Sodium Chloride 2 ml — Single dose 60-90 min preoperatively
  Arms: placebo/sodium chloride

SUMMARY:
The purpose of this study is to evaluate the effect of 125 mg methylprednisolone, given intravenously 60-90 minutes before abdominal surgery,on the postoperative rehabilitation after abdominal hysterectomy.Sodium Chloride is the placebo. The following parameters are registered:

1. Pain 3, 6 and 24 hours postoperatively and 2-7 days after surgery.
2. The postoperative use of additional analgesics.
3. Inflammatory parameters before and after surgery.
4. Time until mobilization.
5. Time until discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients having an abdominal hysterectomy on a benign indication.
* Patients who speak and understand Danish.
* Patients who can give informed consent.

Exclusion Criteria:

* Diabetics
* Regular use of glucocorticoids, opioids or tranquilizers
* Regular treatment with immunosuppressives
* Alcohol or drug abuse
* Morphine intolerance
* Age under 18
* Chronic pain disease eg fibromyalgia, rheumatoid arthritis
* Malign indication for hysterectomy
* BMI over 35
* Decreased kidney function
* ASA III or IV

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pain 6 hours postoperatively | 6 hours postoperatively
  Pain registered by a score on a vas-scale from 0-10 during mobilization and during rest 6 hours postoperatively
Pain 3 hours postoperatively | 3 hours postoperatively
  Pain registered by a score on a vas-scale from 0-10 during mobilization and during rest 3 hours postoperatively
Pain 24 hours postoperatively | 24 hours postoperatively
  Pain registered by a score on a vas-scale from 0-10 during mobilization and during rest 24 hours postoperatively
Pain | 2-7 days postoperatively
  Pain registered by a score on a vas-scale from 0-10 during mobilization and during rest once daily from 2nd-7th postoperative day

SECONDARY OUTCOMES:
Use of additional analgesics | 0-2 days
  The use of other analgesics than paracetamol and diclofenac postoperatively - dosage.
Postoperative nausea | until 2 days postoperatively
  Numbers of vomits
Use of antiemetics | 0-2 days postoperatively
  Dosage of antiemetics during the first 2 days postoperatively
Time until mobilization | 0-2 days
Time until discharge after surgery | 0-10 days
Inflammatory parameters | 0-24 h preoperatively
  CRP measured 0-24 hours preoperatively before injection of project medicine.
Adverse effects | 0-2 days
Inflammatory parameter | 1-2 days postoperative
  CRP measured at 10am on the first and second postoperative day.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Jørgen Secher, Professor, Study Chair — Department of Obstetrics, Hvidovre Hospital
Locations (1):
- Department of Gynaechology and Obstetrics, Holbæk Sygehus, Holbæk, Denmark

REFERENCES:
- [Background] Lidegaard O, Hammerum MS. Landspatientregisteret til kvalitetssikring i det gynækologiske speciale. 2002.
- [Background] Danish hysterektomy database - year report 2004.
- [Background] Hall GM, Peerbhoy D, Shenkin A, Parker CJ, Salmon P. Relationship of the functional recovery after hip arthroplasty to the neuroendocrine and inflammatory responses. Br J Anaesth. 2001 Oct;87(4):537-42. doi: 10.1093/bja/87.4.537. PMID 11878721
- [Background] Henzi I, Walder B, Tramer MR. Dexamethasone for the prevention of postoperative nausea and vomiting: a quantitative systematic review. Anesth Analg. 2000 Jan;90(1):186-94. doi: 10.1097/00000539-200001000-00038. PMID 10625002
- [Background] Wang JJ, Ho ST, Tzeng JI, Tang CS. The effect of timing of dexamethasone administration on its efficacy as a prophylactic antiemetic for postoperative nausea and vomiting. Anesth Analg. 2000 Jul;91(1):136-9. doi: 10.1097/00000539-200007000-00025. PMID 10866900
- [Background] Liu K, Hsu CC, Chia YY. The effective dose of dexamethasone for antiemesis after major gynecological surgery. Anesth Analg. 1999 Nov;89(5):1316-8. PMID 10553859
- [Background] Kehlet H. Glucocorticoids for peri-operative analgesia: how far are we from general recommendations? Acta Anaesthesiol Scand. 2007 Oct;51(9):1133-5. doi: 10.1111/j.1399-6576.2007.01459.x. No abstract available. PMID 17850557
- [Background] Salerno A, Hermann R. Efficacy and safety of steroid use for postoperative pain relief. Update and review of the medical literature. J Bone Joint Surg Am. 2006 Jun;88(6):1361-72. doi: 10.2106/JBJS.D.03018. PMID 16757774
- [Background] Bisgaard T, Klarskov B, Kehlet H, Rosenberg J. Preoperative dexamethasone improves surgical outcome after laparoscopic cholecystectomy: a randomized double-blind placebo-controlled trial. Ann Surg. 2003 Nov;238(5):651-60. doi: 10.1097/01.sla.0000094390.82352.cb. PMID 14578725
- [Background] Romundstad L, Breivik H, Niemi G, Helle A, Stubhaug A. Methylprednisolone intravenously 1 day after surgery has sustained analgesic and opioid-sparing effects. Acta Anaesthesiol Scand. 2004 Nov;48(10):1223-31. doi: 10.1111/j.1399-6576.2004.00480.x. PMID 15504180
- [Background] Nagelschmidt M, Fu ZX, Saad S, Dimmeler S, Neugebauer E. Preoperative high dose methylprednisolone improves patients outcome after abdominal surgery. Eur J Surg. 1999 Oct;165(10):971-8. doi: 10.1080/110241599750008107. PMID 10574107
- [Background] Holte K, Kehlet H. Perioperative single-dose glucocorticoid administration: pathophysiologic effects and clinical implications. J Am Coll Surg. 2002 Nov;195(5):694-712. doi: 10.1016/s1072-7515(02)01491-6. No abstract available. PMID 12437261
- [Background] Sauerland S, Nagelschmidt M, Mallmann P, Neugebauer EA. Risks and benefits of preoperative high dose methylprednisolone in surgical patients: a systematic review. Drug Saf. 2000 Nov;23(5):449-61. doi: 10.2165/00002018-200023050-00007. PMID 11085349
- [Background] Mathiesen O, Rasmussen ML, Dierking G, Lech K, Hilsted KL, Fomsgaard JS, Lose G, Dahl JB. Pregabalin and dexamethasone in combination with paracetamol for postoperative pain control after abdominal hysterectomy. A randomized clinical trial. Acta Anaesthesiol Scand. 2009 Feb;53(2):227-35. doi: 10.1111/j.1399-6576.2008.01821.x. Epub 2008 Dec 6. PMID 19076108
- [Derived] Celik C, Tasdemir N, Abali R, Bastu E, Akbaba E, Yucel SH, Gul A. The effect of uterine straightening by bladder distention before outpatient hysteroscopy: a randomised clinical trial. Eur J Obstet Gynecol Reprod Biol. 2014 Sep;180:89-92. doi: 10.1016/j.ejogrb.2014.06.029. Epub 2014 Jul 7. PMID 25058804
- [Derived] Aabakke AJ, Holst LB, Jorgensen JC, Secher NJ. The effect of a preoperative single-dose methylprednisolone on postoperative pain after abdominal hysterectomy: a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2014 Sep;180:83-8. doi: 10.1016/j.ejogrb.2014.06.026. Epub 2014 Jul 7. PMID 25058803